CLINICAL TRIAL: NCT03681444
Title: Diet Selection Pre-Colonoscopy: Any Difference Between Clear, Low-residue and Regular Diet on Bowel Prep Quality, Tolerance, Acceptance and Compliance
Brief Title: Diet Selection Pre-Colonoscopy: Comparison Between Clear, Low-residue and Regular Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Ghassan Hemadeh, Gastroenterologist, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10218
Record Dates: First submitted 2018-09-19; First posted 2018-09-24 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Bowel Preparation Quality
MeSH Terms: interventions — Diet; Colonoscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular diet (Experimental): no dietary restriction
  Interventions: Other: Regular diet; Diagnostic Test: Colonoscopy
- Clear fluid diet (Placebo Comparator): no solid material
  Interventions: Other: Clear fluid diet; Diagnostic Test: Colonoscopy
- Low residue diet (Experimental): easy digestible food
  Interventions: Other: Low residue diet; Diagnostic Test: Colonoscopy

INTERVENTIONS:
Other: Regular diet — Patients will be provided with any type of food preferred at any time in any quantity
  Arms: Regular diet
Other: Clear fluid diet — Patients will be provided with
  * Plain water
  * Fruit juices without pulp, such as grape juice, filtered apple juice, and cranberry juice
  * Soup broth (bouillon or consommé)
  * Clear sodas, such as ginger ale and Sprite
  * Gelatin (Jell-O)
  * Tea or coffee with no cream or milk added
  * Sports drinks that don't have color
  Arms: Clear fluid diet
Other: Low residue diet — The Low Residue Diet is the same as the soft diet with the added limitation of milk to one pint. It provides foods that are easily digestible. It is often used as a transition diet from liquids to the general diet. Indigestible fiber is reduced by using tender cooked vegetables and ripe, canned or cooked fruits from which the tough skins and seeds have been removed. Tender meat or meat made tender in the cooking process is used, thus reducing the amount of connective tissue.
  Adequacy: By following the recommended guidelines, the diet will be adequate according to the Recommended Daily Allowance.
  Note: For patients with dentures this diet can be modified by the substitution of ground meat for whole meat and excluding all raw vegetables. Personal tolerances determine food choices; avoid foods that cause GI (gastrointestinal) distress prior to the admission even though that food may be on the "foods included" list.
  Arms: Low residue diet
Diagnostic Test: Colonoscopy — Colonoscopy will be performed under conscious sedation with intravenous midazolam and pethidine titrated as required

SUMMARY:
Colonoscopy has been used for ages as an evaluating tool of the colonic mucosa for screening and early detection of colonic cancer. Several studies have reported that poor bowel preparation reduces detection of polyps that may have the potential to be cancerous. Polyethylene glycol (PEG) has become the most commonly used agent for colon cleansing because it does not cause fluid exchange across the mucosal membrane and thereby limits fluid and electrolyte disturbances.

Only a few studies have evaluated the effects of different diet types on bowel preparation under controlled circumstances. Various studies were made to find the best pre-colonoscopy diet with no single clear study comparing all 3 dietary regimen together was carried out. So, evidence for the efficacy of a RD (regular diet) in bowel preparation is lacking, which led us to question whether it is reasonable to recommend a RD for 24 hours prior to colonoscopy as part of a PEG-based bowel prepa¬ration in healthy inpatients.

The investigators are proposing to carry out a randomized clinical trial at Makassed General Hospital and include patients from October 2018 till February 2019. The data of 90 stable adult patients will be obtained through patients' interviews.

In the trial, all adult inpatients (range, 18 to 80 years old) undergoing colonoscopy for colorectal cancer (CRC) screening in Makassed General Hospital with nonspecific gastrointestinal symptoms will be candidates for inclusion in the study. Patient receiving endoscopy will be asked to answer multiple questions on the day of procedure. Patients will be randomly allocated to one of 3 groups: Regular Diet (RD), Clear Fluid (CF) and Low-Residue Diet (LRD). The primary outcome will consist of the quality of bowel preparation and efficacy of colon cleansing.

DETAILED DESCRIPTION:
The study will be conducted in Makassed General Hospital (MGH) including all admitted patients receiving colonoscopy for the different indications. All patients will receive low volume 2L alpha peg split preps given 8 hours apart at a rate of 1 cup q 30 minutes with addition of 1 L of pure water post each liter with the addition 10mg of bisacodyl the night before.

In the trial, all adult inpatients (range, 18 to 80 years old) undergoing colonoscopy for CRC screening In MGH or with nonspecific gastrointestinal symptoms will be candidates for inclusion in the study. Exclusion criteria will be as follows: outpatient status; serious medical condi¬tions, such as severe cardiac, renal, liver, or metabolic disease; stroke or dementia; major psychiatric illness; known allergy to polyethylene glycol (PEG); a previous colon resection; incomplete colonoscopy examination (failure of cecal intubation); or functional constipation defined by Rome III diagnostic criteria.

Patient information was collected before procedure which included age, gender, weight, height, body mass index (BMI), indications for colonoscopy, and history of previous operation and colonoscopy, as well as bowel frequency. Patients will complete a questionnaire before colonoscopy regarding their preparation experience (the start and end time for PEG solution ingestion; the amount of PEG solution ingested; any associated adverse effects, includ¬ing abdominal pain, nausea, vomiting, headache, dizziness, and others; and willingness to repeat the same preparation in the future) with the help of an endoscopy nurse who will be blinded to the dietary randomization.

Participants were categorized into subgroups with regard to compliance; good compliance was defined as less than 25% of the PEG solution remaining, and poor compliance was defined as 25% or more of the PEG solution remaining. The subjects were randomly assigned to either eat Regular diet (RD), clear fluid diet (CLD) or low-residue diet (LRD) explained to each randomized case by in-hospital dietitian. In all three groups the offered diet was given at breakfast and lunch with fluids only given at dinner.

ELIGIBILITY:
Inclusion Criteria:

* inpatients 18 to 75 years old
* undergoing colonoscopy for CRC screening
* with nonspecific gastrointestinal symptoms

Exclusion Criteria:

* outpatient status;
* serious medical conditions, such as severe cardiac, renal, liver, or metabolic disease;
* stroke or dementia;
* major psychiatric illness;
* known allergy to PEG;
* previous colon resection;
* incomplete colonoscopy examination (failure of cecal intubation);
* functional constipation defined by Rome III diagnostic criteria.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
bowel preparation quality: Ottawa bowel preparation scale | within 15 minutes after procedure
  Bowel preparation quality will be assessed by Ottawa bowel preparation scale. The scale assesses three components of the large intestine: (1) the rectosigmoid colon, (2) the mid colon and (3) the right colon.
  A maximum score of 4 is used for each section of the large intestine. A score of 0 is given if the bowel preparation is excellent, a score of 1 is given if the bowel preparation is good, a score of 2 is given if the bowel preparation is fair, a score of 3 is given if the bowel preparation is poor, a score of 4 is given if the bowel preparation is inadequate. The total score is calculated by adding up all 3 scores. The scale has a range from 0 (perfect) to 14 (a completely unprepared colon).

SECONDARY OUTCOMES:
best convenient dietary regimen | before procedure
  Find out the best convenient dietary regimen for pre-colonoscopy preparation evaluated through a questionnaire to assess patient's experience with the bowel preparation model. The questionnaire asks about compliance (good or poor), acceptance (yes or no) and willingness to repeat preparation (yes or no)

CONTACTS AND LOCATIONS:
Overall Officials: Ghassan Hemadeh, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon